CLINICAL TRIAL: NCT03408678
Title: Determinants of Type 2 Diabetes Mellitus Risk in Middle-aged Black South African Men and Women: Dissecting the Role of Sex Hormones, Inflammation and Glucocorticoids
Brief Title: Determinants of Type 2 Diabetes Risk in Middle-aged Black South African Men and Women
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Medical Research Council, South Africa (Other); GlaxoSmithKline (Industry); University of Oxford (Other); University Hospital, Umeå (Other)
Responsible Party: Principal Investigator, Julia Goedecke, Honorary Associate Professor, University of Witwatersrand, South Africa
Other Study IDs: M160604
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Menopause; Hiv
Keywords: body composition; glucocorticoids; inflammation; black African; sex; gonadal steroid hormones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Acquired Immunodeficiency Syndrome; Inflammation; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood retained for extraction of DNA; serum and plasma retained for future biochemical analysis; adipose tissue samples retained for molecular work.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is little known about menopause in African women, whose phenotype differs to Caucasian women, and no data is available on middle-aged black South African men. Accordingly, the study aims to examine the changes in sex hormone levels over the menopausal transition in women, and in men of the same age, and explore the effects on body fat distribution and insulin sensitivity and secretion, dissecting the specific roles of glucocorticoids and inflammatory mediators, in the context of HIV.

Research questions and hypotheses:

1. Does the decrease in sex hormones that occur with ageing increase circulating cortisol and/or inflammatory markers, and directly and/or indirectly via increases in central fat mass, decrease insulin sensitivity in middle-aged black South African men and women?

   Hypothesis: The mechanism underlying the decrease in insulin sensitivity (outcome) associated with the decline in sex hormones (exposure) that occurs with ageing is mediated via an increase in centralization of body fat (mediator), which is due to an increase in inflammation and cortisol production.
2. How does HIV alter the relationship between sex hormones, inflammation and cortisol levels, and subsequently body fat distribution and insulin sensitivity?

   Hypothesis: HIV infection will exacerbate the effects of the decline in sex hormones with ageing, leading to further increases in inflammation and cortisol production, and a consequent increase in the centralization of body fat and decrease in insulin sensitivity.
3. Does adipose tissue glucocorticoid and inflammatory gene expression differ between pre- and post-menopausal women, with and without HIV, and how do these relate to body fat distribution and insulin sensitivity and secretion?

Hypothesis: Adipose tissue estrogen receptor beta (ERβ), 11-beta hydroxysteroid dehydrogenase type 1 (11HSD1) activity and pro-inflammatory markers will be higher in post- compared to pre-menopausal women, which will be exacerbated by HIV infection. This will be associated with down-regulation of subcutaneous adipose tissue (SAT) adipogenic genes, increased visceral adipose tissue (VAT), a decrease in insulin sensitivity and secretion, and consequently an increased risk for type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The study will be performed in two parts:

Part 1 - Using a longitudinal design, a sample of 500 black women at different stages of the menopausal transition, and 500 middle-aged men living in Soweto Johannesburg, South Africa, who were included in previous studies between 2011 and 2014, will be recruited. Socio-demographics, health and menopausal status will be assessed using questionnaires; physical activity and sedentary behaviour will be measured using accelerometry; dietary intake will be estimated using a food frequency questionnaire; body composition and body fat distribution will be assessed using dual energy x-ray absorptiometry (DXA); fasting blood samples will be drawn for the determination of cardio-metabolic risk (glucose, insulin, lipids), cluster of differentiation 4 (CD4) count, as well as sex hormones, inflammatory markers and cortisol concentrations. An oral glucose tolerance test will be performed to measure insulin sensitivity and secretion. Statistical analyses will include multilevel mediation modelling.

Part 2 - Using a cross-sectional design, a sub-sample of 100 women from Part 1 will be selected and divided into four groups including 25 pre-menopausal HIV-negative women and 25 age-matched pre-menopausal HIV-positive women (ARV-Naïve); 25 post-menopausal HIV-negative and 25 age-matched post-menopausal HIV-positive women (ARV-Naïve). The women will undergo a frequently sampled intravenous glucose tolerance test to measure insulin sensitivity and secretion, and adipose tissue biopsies will be taken from the gluteal and abdominal SAT depots for the analysis of gene and protein expression relating to inflammation, sex hormones, glucocorticoid metabolism and adipogenesis. Statistical analyses will include multilevel mediation modelling.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Women on whom baseline data was collected between 2011 and 2014 as part of the Study of Women Entering and in Endocrine Transition.
* Men on whom baseline data was collected in 2014 as part of a larger African genomics study (www.h3Africa.org).

Part 2: A sub-sample of women from Part 1 of the study:

* Pre-menopausal women age-matched within the age range 35-45 years;
* Post-menopausal women age-matched within the age range 55-65 years;
* All women: BMI 25-40 kg/m2

Exclusion Criteria:

Part 1:

- Failed to consent to participate in the study.

Part 2:

* Diabetes, thyroid dysfunction, inflammatory, hepatic and renal diseases;
* Use of hormone replacement therapy; hormonal contraceptives, oral cortisone, anti-inflammatory drugs or antiretroviral therapy;
* Peri-menopausal;
* Currently pregnant or lactating;
* Tobacco use.

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A sample of 500 black women at different stages of the menopausal transition, and 500 middle-aged men living in Soweto Johannesburg, South Africa. The women are a sub-sample of 1007 women on whom baseline data was collected between 2011 and 2014 as part of the Study of Women Entering and in Endocrine Transition. The 500 women will be selected using a random process, to allow their profile to mirror that of the overall sample.
  The men are a sub-sample of 962 black men on whom similar data was collected in 2014 as part of a larger African genomics study (www.h3africa.org). The 500 men will be randomly selected following the same approach applied to the female cohort.
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity and secretion | 4-6 years
  Part 1: insulin sensitivity and secretion estimated from an oral glucose tolerance test; Part 2: insulin sensitivity and secretion estimated using a frequently sampled intravenous glucose tolerance test

SECONDARY OUTCOMES:
Body fat distribution | 4-6 years
  Body fat depots measured using dual energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Julia H Goedecke, PhD, Principal Investigator — Medical Research Council, South Africa; Lisa K Mickelsfield, PhD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- SAMRC/WITS Developmental Pathways of Health Research Unit, University of Witwatersrand, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The principal investigators are prepared to share all individual patient data (IPD) with the wider scientific community, and will make the data available after all the results have been published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication of the data.
Access Criteria: Access will be assessed on a case-by-case basis by the principal investigators of the study.